CLINICAL TRIAL: NCT04277949
Title: Effects of 2,940-nm Fractional Ablative Erbium and Topical DNA Repair Enzymes on p53 Epidermal Expression After 3 Months: A Comparative Clinical Trial
Brief Title: To Evaluate and Compare p53 Epidermal Expression in Healthy Volunteers 3 Months After Treatment With a 2,940-nm Fractional Ablative Erbium Laser and Topical DNA Repair Enzymes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moy-Fincher-Chipps Facial Plastics and Dermatology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 144156
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: p53 Expression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Erbium laser (Experimental): All participants will receive Erbium laser treatment on their right post-auricular region
  Interventions: Device: Erbium:YAG
- DNA repair enzyme (Experimental): All participants will apply topical DNA repair enzymes on their left post-auricular region
  Interventions: Drug: UV endonuclease from Micrococcus luteus

INTERVENTIONS:
Device: Erbium:YAG — Treatment with Erbium:YAG laser
  Arms: Erbium laser
Drug: UV endonuclease from Micrococcus luteus — Application of topical DNA repair enzymes
  Arms: DNA repair enzyme

SUMMARY:
The p53 gene is located on the short arm of chromosome 17 and serves as a tumor suppressor gene. Alteration in p53 is an early event in skin cancer development. Further, p53 is the most commonly mutated gene in non-melanocytic skin cancers. The presence of p53 within epidermal skin cells is believed to reflect the malignant potential of photo-damaged skin. Studies have demonstrated that increasing sun exposure and age are directly associated with higher levels of p53 in facial skin. Consequently, the physiologic overexpression of p53 present in epidermal skin may be indicative of both past photodamage and future risk for developing skin cancer. Advancements in dermatologic research have allowed clinicians to treat photo-damaged skin with with novel modalities. For example, epidermal ablation with the 2,940nm fractional erbium laser has been shown to reduce the risk of carcinogenesis by promoting apoptosis, working similarly to p53. Laser resurfacing results in the replacement of epidermal cells once the necrotic debris is cleared away. This therapeutic effect of laser resurfacing may be gauged by cutaneous p53 expression before and after such interventions. Investigators have noted the reliability of cutaneous p53 expression to gauge therapeutic effects in patients receiving erbium doped yttrium aluminum garnet laser (Er:YAG), dermabrasion, and CO2 laser. Similarly to laser resurfacing, topical DNA repair enzymes have been shown to be protective against skin cancer development and, therefore, may also reduce epidermal p53 expression. UV endonuclease, a DNA repair enzyme derived from the UV-resistant microbe Micrococcus luteus, enhances DNA repair by removing cyclobutane pyrimidine dimers (CPDs) induced by ultraviolet radiation (UVR). To efficiently penetrate the stratum corneum, this enzyme is encapsulated within liposomes, which facilitate entry into keratinocyte nuclei. Once exposed to CPDs, UV endonuclease repairs DNA by catalyzing two reactions: the first uses glycosylase, which releases thymine and causes an apurinic site; the second involves lyase, which incises the phosphodiester backbone, causing a single stranded break. An exonuclease then removes bases around this site, and a polymerase fills the gap, thereby repairing the photodamaged DNA. In addition to repairing damaged DNA on the molecular level, UV endonuclease has also demonstrated the ability to clinically decrease non-melanocytic skin cancer and pre-cancer development. The capability of topical DNA repair enzymes to reverse DNA damage leads us to believe that it will also lead to a reduction in p53 expression within epidermal cells. For these reasons, we wish to investigate the role of 2,940 fractional erbium laser and topical DNA repair enzymes on reducing cutaneous p53 expression.

ELIGIBILITY:
Inclusion Criteria:

* clinical signs of sun damage
* post-auricular regions have been visibly sun exposed

Exclusion Criteria:

* history of actinic keratoses or skin cancer on tested site
* active tanning
* currently taking hormonal replacement therapy
* using topical or oral treatments for for photo aging in previous 6 months
* are currently pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
p53 expression | 3 months
  p53 epidermal expression will be evaluated by scoring the nuclear staining of basilar cells in 3-mm punch biopsies, knowing that the basal layer gives rise to dysplasia. The numbers of stained cells present at the 3-month visit will be compared with the number of stained cells present at the baseline visit.

IPD SHARING:
Plan to Share IPD: No
We are currently in the process of determine the IPD sharing plan

REFERENCES:
- [Background] El-Domyati MB, Attia S, Saleh F, Galaria N, Ahmad H, Gasparro FP, Uitto J. Expression of p53 in normal sun-exposed and protected skin (type IV-V) in different decades of age. Acta Derm Venereol. 2003;83(2):98-104. doi: 10.1080/00015550310007427. PMID 12735636
- [Background] Berg RJ, van Kranen HJ, Rebel HG, de Vries A, van Vloten WA, Van Kreijl CF, van der Leun JC, de Gruijl FR. Early p53 alterations in mouse skin carcinogenesis by UVB radiation: immunohistochemical detection of mutant p53 protein in clusters of preneoplastic epidermal cells. Proc Natl Acad Sci U S A. 1996 Jan 9;93(1):274-8. doi: 10.1073/pnas.93.1.274. PMID 8552621
- [Background] Kanjilal S, Strom SS, Clayman GL, Weber RS, el-Naggar AK, Kapur V, Cummings KK, Hill LA, Spitz MR, Kripke ML, et al. p53 mutations in nonmelanoma skin cancer of the head and neck: molecular evidence for field cancerization. Cancer Res. 1995 Aug 15;55(16):3604-9. PMID 7627969
- [Background] Rees JL. p53 and the origins of skin cancer. J Invest Dermatol. 1995 Jun;104(6):883-4. doi: 10.1111/1523-1747.ep12606149. No abstract available. PMID 7769252
- [Background] Orringer JS, Johnson TM, Kang S, Karimipour DJ, Hammerberg C, Hamilton T, Voorhees JJ, Fisher GJ. Effect of carbon dioxide laser resurfacing on epidermal p53 immunostaining in photodamaged skin. Arch Dermatol. 2004 Sep;140(9):1073-7. doi: 10.1001/archderm.140.9.1073. PMID 15381546
- [Background] Liang SB, Ohtsuki Y, Furihata M, Takeuchi T, Iwata J, Chen BK, Sonobe H. Sun-exposure- and aging-dependent p53 protein accumulation results in growth advantage for tumour cells in carcinogenesis of nonmelanocytic skin cancer. Virchows Arch. 1999 Mar;434(3):193-9. doi: 10.1007/s004280050327. PMID 10190297
- [Background] Borges J, Araujo L, de Oliveira RPB, Manela-Azulay M. Effects of 1,540-nm Fractional Nonablative Erbium and 2,940-nm Fractional Ablative Erbium on p53 Epidermal Expression After 3 months: A Split-Face Interventional Study. Dermatol Surg. 2018 Aug;44(8):1109-1114. doi: 10.1097/DSS.0000000000001527. PMID 29664771
- [Background] El-Domyati MM, Attia SK, Esmat AM, Ahmad HM, Abdel Wahab HM, Badr BM. Effect of laser resurfacing on p53 expression in photoaged facial skin. Dermatol Surg. 2007 Jun;33(6):668-75. doi: 10.1111/j.1524-4725.2007.33141.x. PMID 17550442
- [Background] Kabir Y, Seidel R, Mcknight B, Moy R. DNA repair enzymes: an important role in skin cancer prevention and reversal of photodamage--a review of the literature. J Drugs Dermatol. 2015 Mar;14(3):297-303. PMID 25738852
- [Background] Kuraoka I. Diversity of Endonuclease V: From DNA Repair to RNA Editing. Biomolecules. 2015 Sep 24;5(4):2194-206. doi: 10.3390/biom5042194. PMID 26404388
- [Background] Yarosh D, Klein J, O'Connor A, Hawk J, Rafal E, Wolf P. Effect of topically applied T4 endonuclease V in liposomes on skin cancer in xeroderma pigmentosum: a randomised study. Xeroderma Pigmentosum Study Group. Lancet. 2001 Mar 24;357(9260):926-9. doi: 10.1016/s0140-6736(00)04214-8. PMID 11289350